CLINICAL TRIAL: NCT03554980
Title: Postoperative Pain After Application of Silver Diamine Fluoride Verses Sodium Fluoride Varnish in Treatment of Carious Primary Teeth (A Randomized Clinical Trial)
Brief Title: Application of SDF Verses NaF Varnish in Treatment of Carious Primary Teeth
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa A Salmoon, MSc, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-06-1
Record Dates: First submitted 2018-06-01; First posted 2018-06-13 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Dental Caries in Children
MeSH Terms: interventions — silver diamine fluoride; Bifluorid 12

STUDY DESIGN:
Intervention Model Description: patient will receive either Silver Diamine Fluoride or Sodium Fluoride varnish according to the allocation ratio
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1 (Experimental): 38% silver diamine fluoride liquid will be applied twice annually and patients will be followed up at 0,1,3,6, 9 and 12.
  SDF is a brush-on liquid.
  Interventions: Drug: Silver Diamine Fluoride
- Group 2 (Active Comparator): 5% sodium fluoride varnish will be applied four times annually and patients will be followed up at 0,1,3,6,9 and 12.
  Interventions: Drug: Sodium Fluoride varnish

INTERVENTIONS:
Drug: Silver Diamine Fluoride — SDF will be applied with a brush.
  Other Names: SDF
  Arms: Group 1
Drug: Sodium Fluoride varnish — NaF will be applied with a brush
  Other Names: NaF varnish
  Arms: Group 2

SUMMARY:
The aim of this study is to assess the postoperative pain after application of silver diamine fluoride versus sodium fluoride varnish in treatment of carious primary teeth.

DETAILED DESCRIPTION:
Untreated dental decay and poor access to dental care are significant Public health problems for children in the world (Dye et al. 2015 and Horst, 2016). Early childhood caries is a multifactorial, infectious and transmissible dental disease affecting young children . Conventional restorative treatment may fail to reduce the burden of early childhood caries in many parts of the world. Most decayed teeth in preschool children remained unrestored . Consequences of untreated decay in preschool children may include increased risk of future caries in primary and permanent dentition, pain and infections; increased expensive emergency room visits and hospital admissions; increased treatment costs because of extensive decay and the accompanying need for general anesthesia; delayed growth and development; and missed days from school and work .To reduce the burden of caries disease in young children and to avoid possible serious consequences of untreated decay, it is important to identify an effective, low-cost method of treating caries in children at high risk of caries and with limited access to dental care. Silver diamine fluoride (SDF) has been identified as an anticariogenic agent that successfully arrests dental decay and has the potential to address the epidemic of untreated decay in young children

Therefore this study will be conducted to assess the postoperative pain after application of silver diamine fluoride versus sodium fluoride varnish in treatment of carious primary teeth.

Benefits of the research to the patient:

According to American Academy of Pediatric Dentistry (AAPD), 2017 SDF application is:

* Safe.
* Noninvasive.
* Inexpensive.
* Effective in dental caries management, especially arresting cavitated caries lesions in the primary dentition.

Benefits of the research to the clinician:

According to AAPD, 2017 SDF is:

* Easily performed.
* A promising strategy to manage dental caries in very young children or those who have special needs.
* Doesn't require cooperation from children during dental treatment.

It will improve patient confidence with the dentist

Explanation for choice of comparators:

The use of sodium fluoride is well documented in the literature as successful caries arrestment material. Arrestment proportion of caries for sodium fluoride varnish was found to be 84.4% (NaF) and 85.3% for ( NaF + chlorohexidine mouth wash) .

ELIGIBILITY:
Inclusion Criteria:

1. Children with carious primary teeth before eruption of permanent teeth
2. High caries risk patients with anterior or posterior carious lesions.
3. Uncooperative children without access to or with difficulty accessing dental care.

Exclusion Criteria:

1. Children with spontaneous or elicited pain from caries
2. Tooth mobility
3. Signs of pulpal infection
4. Severe medical conditions that would not allow management in the clinic
5. Hereditary developmental defects, such as amelogenesis imperfecta or dentinogenesis imperfecta
6. Known allergies or sensitivities to dental materials, including SDF
7. Inability to return for recall visits
8. Refusal of participation from the guardian or parents

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain | 12 months
  Postoperative pain will be assessed through questioning the patient and/or parent .Binary (Yes or No)

SECONDARY OUTCOMES:
Parental satisfaction | 12 months
  Parental satisfaction will be assessed through questioning the parent. Binary (yes or no)
Caries arrest (dentin texture) Cries arrest (Dentine texture) | 12 months
  Caries arrest will be assessed through tactile examination (hard or soft). Categorical
Discoloration (yellow, brown, black) | 12 months
  Discoloration will be assessed through visual examination. Categorical

CONTACTS AND LOCATIONS:
Overall Officials: Nevine G Waly, Professor, Study Chair — Pediatric Dentistry, Faculty of Dentistry, Cairo University; Eman S Elmasry, Professor, Study Director — Pediatric Dentistry, Faculty of Dentistry, Cairo University; Fatma KI Abdelgawad, Lecturer, Study Director — Pediatric Dentistry, Faculty of Dentistry, Cairo University; Marwa A Salmoon, MSc, Principal Investigator — Pediatric Dentistry, Faculty of Dentistry, Cairo University
Locations (1):
- Pediatric Dentistry, Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
outcome results for both groups will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: to be determined later
Access Criteria: to be determined later